CLINICAL TRIAL: NCT06058715
Title: TAP Block Versus Conventional Systemic Analgesia in Laparoscopic Surgery: A Prospective Randomized Trial
Brief Title: TAP Block Versus Conventional Systemic Analgesia
Acronym: TAPLAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Scientific Research, Tunisia (Other Government)
Responsible Party: Principal Investigator, Sana Landolsi, Associate professor in general surgery, University Tunis El Manar, Faculty of medicine of Tunis, Department of surgery, Mahmoud El Matri hospital, Ariana, Tunisia, Ministry of Scientific Research, Tunisia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAP1-LAP2
Record Dates: First submitted 2023-06-08; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block (Experimental): Bilateral TAP block is administered intraoperatively at laparoscopy, directly after insufflation and insertion of the first trocar and camera. The ultrasound probe is placed longitudinally on the midaxillary line near umbilicus, and the transversus abdominis and internal oblique muscles are scanned and observed. The needle (22-gauge 90 mm disposable spinal needle) is inserted in plane. After placing the needle-tip into the fascia between transversus abdominis and internal oblique muscles, Ropivacaine 0.25% (Naropin) is injected bilaterally at the dose of 0.5 mg/kg. It is all done by one Anesthetist which is expert in that area and is not in charge of collecting the data.
  No additional regional anesthesia, including epidural or spinal anesthesia, is given.
  The patients are mobilized in the recovery room 2 h after surgery.
  Interventions: Procedure: Transverse Abdominal Plan block (TAP block)
- Conventional analgesia (Active Comparator): No additional regional anesthesia, including epidural or spinal anesthesia, is given.
  For postoperative analgesia, all patients receive paracetamol intravenously at the dose of 1 g three times up to 24 hours, starting immediately after surgery. Complementary opioids are given on request when pain numerical rating scale (pain NRS) : NRS > 3 at rest or for pain NRS > 5 on exercise. Oxycodone is given intravenously at the dose of 0.05 mg/kg only in the recovery room up to two hours after the surgery. It is administrated intramuscularly at the dose of 0.1 mg/kg up to 24 hours after surgery. Then, it is given orally at the dose of 0.2 mg/kg from 24 to 48 hours after surgery.
  Interventions: Procedure: Transverse Abdominal Plan block (TAP block)

INTERVENTIONS:
Procedure: Transverse Abdominal Plan block (TAP block) — Bilateral TAP block is administered intraoperatively at laparoscopy, directly after insufflation and insertion of the first trocar and camera. The ultrasound probe is placed longitudinally on the midaxillary line near umbilicus, and the transversus abdominis and internal oblique muscles are scanned and observed. The needle (22-gauge 90 mm disposable spinal needle) is inserted in plane and after placing the needle-tip into the fascia between transversus abdominis and internal oblique muscles, 20 ml of ropivacaine 0.25% is injected bilaterally. It is all done by one Anesthetist which is expert in that area and is not in charge of collecting the data.

SUMMARY:
The goal of this clinical trial is to compare TAP block to conventional systemic analgesia for postoperative pain management in patients undergoing elective laparoscopic cholecystectomy. As the adverse effects of pain management is related to size of opioid dose use, opioid consumption is chosen as the primary outcome and a decrease of at least 20% in the TAP block compared with the conventional systemic analgesia is considered to be clinically significant.

Written informed consent has to obtained from all study patients. This trial is a prospective parallel group randomized superiority trial comparing TAP block to classic systemic analgesia in patients undergoing elective laparoscopic surgery in the department of surgery, Mahmoud El Matri Hospital, Ariana, with a 1:1 allocation ratio.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy constitutes a routinely performed procedure world-wide. Analgesia accounts for one of the major keys for success especially in enhanced recovery after surgery pathway and ambulatory surgery. Hence, controlling opioid consumption used in conventional systemic analgesia is mandatory while reliving pain. The TAP block is integrated within a multimodal analgesia. It corresponds to a locoregional analgesia.

The goal of this clinical trial is to compare TAP block to conventional systemic analgesia for postoperative pain management in patients undergoing elective laparoscopic cholecystectomy. As the adverse effects of pain management is related to size of opioid dose use, opioid consumption is chosen as the primary outcome and a decrease of at least 20% in the TAP block compared with the conventional systemic analgesia is considered to be clinically significant.

Written informed consent has to obtained from all study patients. This trial is a prospective parallel group randomized superiority trial comparing TAP block to classic systemic analgesia in patients undergoing elective laparoscopic surgery in the department of surgery, Mahmoud El Matri Hospital, Ariana, with a 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

All patients scheduled for elective laparoscopic cholecystectomy at the department of surgery, Mahmoud El Matri Hospital, Ariana

Exclusion Criteria:

* Severe renal insufficiency (GFR < 30 ml/min)
* Severe hepatic insufficiency (TT ≤ 50%)
* Severe COPD (FEV1 > 30%)
* Metastatic malignancy
* Hematologic disease or a congenital clotting disorder
* Preoperative opioid use
* Age under 18 years
* Pregnancy or breast-feeding
* Hyper-reactivity toward ropivacaine
* Estimated risk for conversion to open surgery > 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption during the first 48 h postoperatively. | Every six hours
  Opioids are given only on request based on pain numerical rating scale (pain NRS) varying from 0 to10. For pain NRS > 3 at rest or for pain NRS > 5 on exercise, oxycodone is administrated intravenously at the recovery room at the dose of 0.05 mg/kg. Then, it is used intramuscularly at the dose of 0.1 mg/kg up to 24 hours after surgery and orally at the dose of 0.15 mg/kg between 24 and 48 hours after surgery.
  At 2 to 4 weeks postoperatively, all patients are contacted either by phone or at the outpatient clinic during a follow-up visit and asked to complete a form with questions evaluating pain sensations, pain intensity, need for pain medication, performance of daily activities, and any limitations of these due to postoperative abdominal pain.

SECONDARY OUTCOMES:
Pain intensity on a numerical rating scale (pain NRS, 0-10) | Every six hours
  pain intensity is measured 30 min after arrival and then every hour until the patient is discharged to the ward. In the ward, the pain NRS score is measured for each consecutive 6-h block. Means of the first and second 6-h blocks and third and fourth blocks are calculated and used for further analysis. Additionally, the maximal daily pain NRS scores are collected. At the time of discharge, patients evaluate their satisfaction with pain management as a whole (scale 0-3: 0 poor; 3 excellent).
Postoperative evaluation at 4 weeks | At 4 weeks after surgery
  At 4 weeks postoperatively, all patients are contacted either by phone and asked to complete a form with questions evaluating pain sensations, pain intensity, need for pain medication, performance of daily activities, and any limitations of these due to postoperative abdominal pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of surgery, Mahmoud El Matri hospital, Ariana, Tunisia, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: No